CLINICAL TRIAL: NCT06060158
Title: Feasibility of Internet-Delivered Group Cognitive Behavioral Therapy for Insomnia in Gynecologic Oncology Patients
Brief Title: Feasibility of Internet Group CBT-I for Gyn Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1636910
Record Dates: First submitted 2023-06-29; First posted 2023-09-29 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility study looking at delivering small group therapy online.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT-I online group (Experimental): Twelve eligible participants will meet weekly for 6 weeks while undergoing the CBT-I program. At the end of each weekly session, participants will complete a survey reviewing the acceptability of undergoing insomnia treatment in an internet-based small-group setting.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — 6 sessions

SUMMARY:
The goal of this study is to evaluate the feasibility and acceptability of delivering cognitive behavioral therapy for insomnia (CBT-I) to gynecologic cancer patients in an internet-based small-group setting.

Secondary objectives:

1. To compare insomnia symptoms before and after intervention.
2. To evaluate any changes in quality of life symptoms while undergoing the intervention.
3. To evaluate the duration of symptoms improvement after the intervention is complete.

DETAILED DESCRIPTION:
This is a pilot feasibility study looking at delivering CBT-I to gynecologic cancer patients. This study will be completed via a novel internet based small group platform. Twelve eligible participants will meet weekly for 6 weeks while undergoing the CBT-I program.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking women greater than 18 years old who present to UC Davis Comprehensive Cancer Center for treatment or surveillance of gynecologic cancer
2. Must have access to internet
3. Be able to connect via secure web-based platform
4. Be able to complete online questionnaires
5. Moderate or severe insomnia
6. Have access to a mobile device or computer

Exclusion Criteria:

1. Participants without ability to connect with both audio and visual through secure web-based platform
2. Participant is currently taking sleep medication prescribed by their provider for sleep disturbance or insomnia - Patients taking over the counter medications or supplements are eligible
3. Participants with remote history of insomnia, but not currently having symptoms of insomnia
4. Have other reasons for poor sleep

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Attendance | 6 weeks
  Main feasibility metric, recorded as number of sessions successfully attended. Participants would need to attend at least 4 sessions of the CBT-I sessions. Therefore, attendance among all participants must be 67% or greater to be considered feasible. A session must be attended for at least 50% of the time or will be counted as missed.
Acceptability | 24 weeks
  A three-question survey at the end of each session. Question 1 is yes/no, questions 2 and 3 are write in. At the end of the program, a longer acceptability survey will be conducted. If a participant's response to question 1 indicates acceptability for a given session, that session will be deemed 'acceptable'. If 50% or more of participants rated the session as acceptable, then that session will be rated as acceptable.

SECONDARY OUTCOMES:
Insomnia symptoms | 24 weeks
  Measured by Insomnia Severity Index (ISI) with scale range of 0 to 27, higher numbers indicating more severe insomnia
Changes in quality of life symptoms | 24 weeks
  Measured by the 7-item Functional Assessment of Cancer Therapy (FACT-G7) Assessment, with likhert scales from 0-4 and higher numbers indicating more severe symptoms
Sleep Quality | 24 weeks
  Measured by the Pittsburgh Sleep Quality Index (PSQI), score of 0-21 points, higher score indicating more severe difficulty sleeping.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chen, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No